CLINICAL TRIAL: NCT03861611
Title: A Comparison of NSAIDs for Acute, Non-radicular Low Back Pain. A Randomized Trial
Brief Title: A Comparison of NSAIDs for Acute, Non-radicular Low Back Pain.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Eddie Irizarry, Assistant Professor of Emergency Medicine, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-10026
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Results first posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Back Pain Without Radiation; Low Back Pain
Keywords: ketorolac; diclofenac; ibuprofen; low back pain; back pain
MeSH Terms: conditions — Back Pain; Low Back Pain | interventions — Ketorolac; Ibuprofen; Diclofenac; Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ketorolac + Educational Intervention (Experimental): Participants may be randomized to receive Ketorolac for their LBP. Research personnel will provide each participant with a 15-minute educational intervention.
  Interventions: Drug: Ketorolac; Behavioral: Educational Intervention
- Ibuprofen + Educational Intervention (Experimental): Participants may be randomized to receive Ibuprofen for their LBP. Research personnel will provide each participant with a 15-minute educational intervention.
  Interventions: Drug: Ibuprofen; Behavioral: Educational Intervention
- Diclofenac + Educational Intervention (Experimental): Participants may be randomized to receive diclofenac for their LBP. Research personnel will provide each participant with a 15-minute educational intervention.
  Interventions: Drug: Diclofenac; Behavioral: Educational Intervention

INTERVENTIONS:
Drug: Ketorolac — Participants may be randomized to receive Ketorolac oral medication 10 mg, every 8 hours for 5 days as needed
  Arms: Ketorolac + Educational Intervention
Drug: Ibuprofen — Participants may be randomized to receive Ibuprofen oral medication 600 mg, every 8 hours for 5 days as needed
  Arms: Ibuprofen + Educational Intervention
Drug: Diclofenac — Participants may be randomized to receive Diflofenac oral medication 50 mg, every 8 hours for 5 days as needed
  Arms: Diclofenac + Educational Intervention
Behavioral: Educational Intervention — Research personnel will provide each patient with a 15-minute educational intervention. This will be based on National Institute of Arthritis and Musculoskeletal and Skin Diseases Handout on Health: Back Pain information

SUMMARY:
Purpose: This is a randomized clinical trial comparing the effects of three different medications for acute low back pain (LBP):Ketorolac, Ibuprofen, Diclofenac

Hypothesis: A daily regimen of ketorolac will provide greater relief of LBP than ibuprofen or diclofenac 5 days after an emergency department (ED) visit, as measured by the Roland Morris Disability Questionnaire (RMQ)

DETAILED DESCRIPTION:
More than 2.5 million patients present to US emergency departments (ED) annually with low back pain. Up to half of ED patients with acute, new onset low back pain (LBP) report persistent moderate or severe pain one week after the ED visit. Non-steroidal anti-inflammatory drugs (NSAIDs) are an effective treatment of acute LBP, though their impact is only modest.Given the poor pain and functional outcomes that persist beyond an ED visit for acute LBP, this clinical trial proposes to determine whether there is a difference in efficacy between the NSAIDs ketorolac, ibuprofen, and diclofenac and for the treatment of acute, non-traumatic, non-radicular low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age 18-64.
* Present to ED primary for management of Low Back Pain (LBP)
* Functionally impairing back pain: A baseline score of greater than 5 on the Roland-Morris Disability Questionnaire
* Musculoskeletal etiology of low back.
* Non-radicular pain.
* Pain duration <2 weeks (336 hours).
* Non-traumatic LBP
* Participant is to be discharged home.

Exclusion Criteria:

* Flank pain, that is pain originating from tissues lateral to the paraspinal muscles.
* Not available for follow-up
* Pregnant
* Chronic pain syndrome
* Allergic to or intolerant of investigational medications
* Contra-indications to investigational medications

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eddie Irizarry, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share

REFERENCES:
- See also: National Institute of Arthritis and Musculoskeletal and Skin Diseases Handout on Health: Back Pain information — http://www.niams.nih.gov/Health_Info/Back_Pain/default.asp

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketorolac + Educational Intervention: Participants may be randomized to receive Ketorolac for their LBP. Research personnel will provide each participant with a 15-minute educational intervention.
  Ketorolac: Participants may be randomized to receive Ketorolac oral medication 10 mg, every 8 hours for 5 days as needed
  Educational Intervention: Research personnel will provide each patient with a 15-minute educational intervention. This will be based on National Institute of Arthritis and Musculoskeletal and Skin Diseases Handout on Health: Back Pain information webpage
- Ibuprofen + Educational Intervention: Participants may be randomized to receive Ibuprofen for their LBP. Research personnel will provide each participant with a 15-minute educational intervention.
  Ibuprofen: Participants may be randomized to receive Ibuprofen oral medication 600 mg, every 8 hours for 5 days as needed
  Educational Intervention: Research personnel will provide each patient with a 15-minute educational intervention. This will be based on National Institute of Arthritis and Musculoskeletal and Skin Diseases Handout on Health: Back Pain information webpage
- Diclofenac + Educational Intervention: Participants may be randomized to receive diclofenac for their LBP. Research personnel will provide each participant with a 15-minute educational intervention.
  Diclofenac: Participants may be randomized to receive Diclofenac oral medication 50 mg, every 8 hours for 5 days as needed
  Educational Intervention: Research personnel will provide each patient with a 15-minute educational intervention. This will be based on National Institute of Arthritis and Musculoskeletal and Skin Diseases Handout on Health: Back Pain information webpage
Period: Overall Study
Arm/Group | Ketorolac + Educational Intervention | Ibuprofen + Educational Intervention | Diclofenac + Educational Intervention
Started | 66 | 66 | 66
Completed | 59 | 61 | 62
Not Completed | 7 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Ketorolac + Educational Intervention: Participants may be randomized to receive Ketorolac for their LBP. Research personnel will provide each participant with a 15-minute educational intervention.
  Ketorolac: Participants may be randomized to receive Ketorolac oral medication 10 mg, every 8 hours for 5 days as needed
  Educational Intervention: Research personnel will provide each patient with a 15-minute educational intervention. This will be based on National Institute of Arthritis and Musculoskeletal and Skin Diseases Handout on Health: Back Pain information webpage (available at http://www.niams.nih.gov/Health_Info/Back_Pain/default.asp)
- Ibuprofen + Educational Intervention: Participants may be randomized to receive Ibuprofen for their LBP. Research personnel will provide each participant with a 15-minute educational intervention.
  Ibuprofen: Participants may be randomized to receive Ibuprofen oral medication 600 mg, every 8 hours for 5 days as needed
  Educational Intervention: Research personnel will provide each patient with a 15-minute educational intervention. This will be based on National Institute of Arthritis and Musculoskeletal and Skin Diseases Handout on Health: Back Pain information webpage (available at http://www.niams.nih.gov/Health_Info/Back_Pain/default.asp)
- Diclofenac + Educational Intervention: Participants may be randomized to receive diclofenac for their LBP. Research personnel will provide each participant with a 15-minute educational intervention.
  Diclofenac: Participants may be randomized to receive Diclofenac oral medication 50 mg, every 8 hours for 5 days as needed
  Educational Intervention: Research personnel will provide each patient with a 15-minute educational intervention. This will be based on National Institute of Arthritis and Musculoskeletal and Skin Diseases Handout on Health: Back Pain information webpage (available at http://www.niams.nih.gov/Health_Info/Back_Pain/default.asp)
- Total: Total of all reporting groups
Arm/Group | Ketorolac + Educational Intervention | Ibuprofen + Educational Intervention | Diclofenac + Educational Intervention | Total
Number analyzed (Participants) | 66 | 66 | 66 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (11.2) | 40.3 (11.4) | 39.9 (10.1) | 39.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 25 | 74
  Male | 41 | 42 | 41 | 124
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 5 in Functional Impairment
Description: The change will be assessed by Roland Morris Disability Questionnaire between the baseline ED visit and the five day follow-up. The Roland-Morris Questionnaire (RMQ) is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale (0-24).
Time Frame: Baseline to 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketorolac + Educational Intervention | Ibuprofen + Educational Intervention | Diclofenac + Educational Intervention
Number analyzed (Participants) | 59 | 61 | 62
score on a scale | 11.9 (8.8) | 9.4 (9.5) | 10.9 (9.4)

2. Secondary Outcome: Worst LBP 2 Days After ED Visit
Description: Participants were called 2 days after ED visit and asked to report their worst LBP experienced over the previous 24 hours, using a four point ordinal scale: severe, moderate, mild, or none.
Time Frame: 2 days after Emergency department visit
Population: Participants with missing data not reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac + Educational Intervention | Ibuprofen + Educational Intervention | Diclofenac + Educational Intervention
Number analyzed (Participants) | 61 | 62 | 63
Participants
  None | 8 | 10 | 13
  Mild | 29 | 18 | 25
  Moderate | 18 | 23 | 18
  Severe | 6 | 11 | 7

3. Secondary Outcome: Frequency of LBP 2 Days After ED Visit
Description: Participants were called 2 days after ED visit and asked to report the frequency of LBP experienced over the previous 24 hours. Frequency was assessed using the five point Likert scale: Not at all, Rarely, Sometimes, Usually, Always
Time Frame: 2 days after Emergency department visit
Population: Participants with missing data not reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac + Educational Intervention | Ibuprofen + Educational Intervention | Diclofenac + Educational Intervention
Number analyzed (Participants) | 61 | 62 | 63
Participants
  Never | 6 | 7 | 10
  Rarely | 18 | 10 | 14
  Sometimes | 26 | 21 | 21
  Frequently | 5 | 9 | 7
  Always | 6 | 15 | 11

4. Secondary Outcome: How Often Participants Used Assigned Medication
Time Frame: 24 hours to 5 days
Population: Participants with missing data not reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac + Educational Intervention | Ibuprofen + Educational Intervention | Diclofenac + Educational Intervention
Number analyzed (Participants) | 59 | 61 | 63
Participants
  Never | 2 | 1 | 0
  Only Once | 3 | 5 | 3
  Sometimes | 10 | 4 | 7
  Once a day | 26 | 18 | 15
  Twice or more a day | 18 | 33 | 38

ADVERSE EVENTS:
Time Frame: 5 days
Description: Study participants were asked: Did you have any side effects from the medications you've been taking for low back pain? Study participants were also asked: Did the medication irritate your stomach? 1 patient randomized to ibuprofen was admitted to the hospital for angioedema which was may have been due to concomitant angiotensin converting enzyme inhibitor use.
Arm/Group | Ketorolac + Educational Intervention | Ibuprofen + Educational Intervention | Diclofenac + Educational Intervention
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 1/66 | 0/66
Other Adverse Events (participants affected / at risk) | 3/66 | 16/66 | 6/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac + Educational Intervention (N=66) | Ibuprofen + Educational Intervention (N=66) | Diclofenac + Educational Intervention (N=66)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — One participant in the ibuprofen arm was admitted to the hospital for angioedema. This participant was taking an angiotensin converting enzyme inhibitor, which was thought to be the more likely cause of this clinical presentation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ketorolac + Educational Intervention (N=66) | Ibuprofen + Educational Intervention (N=66) | Diclofenac + Educational Intervention (N=66)
Stomach irritation (Gastrointestinal disorders) | 3 | 16 | 6 — Study participants were asked: Did the medication irritate your stomach?

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT03861611/Prot_SAP_000.pdf